CLINICAL TRIAL: NCT06775223
Title: Assessment of Validity and Reliability of the Turkish Version of the Quality of Life and Related Events Assessment Scale for Pacemaker Patients
Status: Recruiting | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gamze Nur AHISKALI, Physiotherapist Gamze Nur AHISKALI, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2024-29
Record Dates: First submitted 2024-09-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Implantable Electronic Devices; Quality of Life
Keywords: quality of life; patient reported outcomes; cardiac implantable electronic devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac implantable electronic devices — validity and reliability study

SUMMARY:
Cardiac implantable electronic devices are widely utilized to lower the rates of morbidity and mortality from ventricular tachycardia and ventricular fibrillation, as well as the incidence of sudden cardiac death. Although implantation of these devices increases survival rates, patients may experience acute and chronic complications. These complications include device dislocation and fracture, inappropriate shocks, pocket hematoma, or infection. Furthermore, functional loss in the upper extremity may result from upper extremity restrictions that are applied for an excessively long time in order to ensure proper placement of the device following implantation, or from patients who choose to extend this period on their own initiative out of worry about device failure or dislocation. Patients' quality of life may be negatively impacted by these issues as well as diminished exercise capacity, weariness, and weaker respiratory and peripheral muscles. A quality of life scale called 'The Assessment of Quality of Life and Related Events (AQUAREL)' was developed by Stoffmel et al. for patients using pacemakers. In this study, the validity and reliability study of the Turkish version of the AQAREL Scale will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Having a pacemaker implant and not having any complications at the last pacemaker check-up,

  * Being in NYHA I-II-III-IV class,
  * Patients with no cooperation problems,
  * Volunteering to participate in the study.

Exclusion Criteria:

* • Patients with insufficient dementia or cognitive impairment due to multiple comorbidities (e.g., recent cerebrovascular accident and/or significant hypotension),

  * Patients with a history of psychiatric illness,
  * Patients with speech, hearing or intellectual disabilities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participant with cardiac implantable electronic devices between the ages of 18-65
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Turkish adaptation of the scale assessing quality of life | 1 years
  The Assessment of Quality of Life And RELated Events (AQUAREL) scale, which was created especially for people with cardiac implanted electronic devices, will be translated into Turkish. / The total score ranges from 0 to 100. A low score reflects poor health perception, loss of function and presence of pain, while a high score reflects good health perception, preserved function and absence of pain.

SECONDARY OUTCOMES:
Evaluation of quality of life | 1 year
  Short Form- 36 -SF-36 Life Questionnaire / Each sub-parameter is scored between 0 and 100. A high score indicates that the individual has a high quality of life.
Evaluation of quality of life | 1 year
  MacNew Heart Disease Health-Related Quality of Life Questionnaire / The questions are scored from 1 to 7, with higher scores indicating better quality of life.
Evaluation of activities of daily living | 1 year
  Performance Measure for Activities of Daily Living-8 for Patient with Mild Symptomatic Heart Failure- PMADL-8 / The total score ranges from 8-32, with a high score indicating a level of limitation in activities of daily living.
Evaluation of comorbidity level | 1 year
  Modified Charlson Comorbidity İndex (CCI) / Comorbidity classification is low (score ≤ 3), moderate (score 4 and 5), high (score 6 and 7) and very high comorbidity (score ≥ 8). High score indicates high mortality rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Corum Erol Olçok Training and Research Hospital, Çorum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No